CLINICAL TRIAL: NCT06113796
Title: Economic Analysis of Robotic Rectal Resection in German Health Care System
Status: Completed | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Other Study IDs: UKE Hamburg 3
Record Dates: First submitted 2023-10-04; First posted 2023-11-02 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-11

CONDITIONS: Rectal Cancer
Keywords: Robotic Surgery; Rectal Cancer; Low anterior Resection; Abdominoperineal rectal extirpation; Economic analysis
MeSH Terms: conditions — Rectal Neoplasms | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Robotic sphincter-preserving rectal resection: Patients with robotic anterior or low anterior rectal resection and primary anastomosis for rectal cancer.
  Interventions: Other: Surgery
- Robotic abdominoperineal rectal resection: Patients with robotic abdominoperineal rectal resection for rectal cancer.
  Interventions: Other: Surgery

INTERVENTIONS:
Other: Surgery — Robotic rectal resection, either sphincter preserving or extirpation

SUMMARY:
Analysis of cost effectiveness of robotic rectal resection, either sphincter preserving or abdominoperineal extirpation, in the German diagnosis related groups (DRG) system.

DETAILED DESCRIPTION:
Robotic surgery has many well-known benefits for patients and surgeons, while it comes with higher acquisition and maintenance costs. On the other hand, a higher proportion of minimally invasive procedures can save costs by reducing complications, decreasing hospital stays due to lower morbidity, and saving personnel.

To what extent can robotic surgery be cost-covering or even profitable, depending on the postoperative course? This question is investigated under the conditions of the German DRG system.

ELIGIBILITY:
Inclusion Criteria:

* 18y
* histologically proven rectal cancer with curative therapeutic approach
* suitable for minimally-invasive surgery

Exclusion Criteria:

* no rectal cancer
* primary open surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients operated robotically-assisted between 01/2018 and 12/2019 for rectal cancer are suitable for inclusion.
Sampling Method: Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Costs of treatment | 1 year
  costs caused by the case

SECONDARY OUTCOMES:
Major Complication | 30 days postoperatively
  Clavin Dindo Score ≥ 3
Length of Hospital Stay | 3 months
  Hospital Stay after Surgery
30-days Readmission | 30 days
  Readmission within 30 days after Surgery

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Perez, Prof., Principal Investigator — Department of General, Visceral and Thoracic Surgery, University Hospital Hamburg-Eppendorf
Locations (1):
- University of Hamburg Medical Institutions, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No